CLINICAL TRIAL: NCT04023851
Title: Mobile Application of Seizure Diary (Brain4U) in Epilepsy for the Better Patient Care
Brief Title: Mobile Application of Seizure Diary (Brain4U) in Epilepsy Care
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hunmin Kim, Associate Professor, Seoul National University Hospital
Other Study IDs: 01
Record Dates: First submitted 2019-07-15; First posted 2019-07-18 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Epilepsy
Keywords: Epilepsy; Seizure diary; Mobile application
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adolescent patient: * Participant between the ages of 15-18
  * Participants who are taking antiepileptic drug for seizure control
  Interventions: Device: Mobile application Brain4U
- Parents with epilepsy children: * Participants who have child with epilepsy (ages of 1-15)
  * Participants' child who are taking antiepileptic drug for seizure control
  Interventions: Device: Mobile application Brain4U

INTERVENTIONS:
Device: Mobile application Brain4U — Brain4U application provides participants to record seizures, medications, side effects, and combined psychiatric problems. It also reminds participants when to take antiepileptic drugs.

SUMMARY:
The study is intended to evaluate the impact of mobile application on management and knowledge acquisition in patients with epilepsy.

DETAILED DESCRIPTION:
Investigators assess the general and personal knowledge of epilepsy, compliance of antiepileptic drugs (AED), and self efficacy scale. Participants be asked to use the mobile application (Brain4U) and record seizure type, frequency of seizures, aggravating factors, and adverse events related to antiepileptic drugs for 2 month period.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between the ages of 1-99.
* Participants must attend Seoul National University Bundang Hospital Pediatric Neurology Outpatient Clinic.
* Participants under age 18 must have an adult guardian give informed consent.
* Participants must have a functioning smartphone (iOS or Android) which can download the and perform Brain4U application.
* Participants must be able to use mobile application skillfully.

Exclusion Criteria:

* Person who does not have smartphone nor restricted to use mobile application can not participate this study.
* Person with intellectual disability or unable to use mobile application can not participate this study.

Ages: 1 Year to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: There are 2 groups of study population in this study:
  Adolescent patients with epilepsy and Parents with epilepsy children.
  1. Adolescent patient
     * Participant between the ages of 15-18
     * Participants who are taking antiepileptic drug for seizure control
  2. Parents with epilepsy children
     * Participants who have child with epilepsy (ages of 1-15)
     * Participants' child who are taking antiepileptic drug for seizure control
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of knowledge acquisition in epilepsy | 2 months
  Baseline and 2 month Timepoint scores from questionnaires are assessed. Improvement in knowledge acquisition and self-efficacy by using questionnaire.
  1. Genetal knowledge (G) Questionnaire:
     There are total 10 questions (1 point score for each question) to evaluate general knowlege about epilepsy.
     Score reported as (mean, SD), higher scores are better. Score ranges 0 to 10.
  2. Persional knowledge (P) questionnaire:
     There are total 4 questions (1 point score for each question) to evaluate knowlege about individual's epilepsy.
     Score reported as (mean, SD), higher scores are better. Score ranges 0 to 4.
  3. Self-efficacy scale (SE): There are 4 questions (1 point score for each question) to evaluate self-efficacy scale.
  Score reported as (mean, SD), higher scores are better. Score ranges 0 to 4.

SECONDARY OUTCOMES:
AED compliance | 2 months
  Baseline and 2 month Timepoint AED compliances are reported.
  Assess improvement of AED compliance by comparing "Days with AED per month" before and after using mobile application.
  Count the "Days with AED" in a month and converted to the percentage.
  Percentage ranges 0 to 100%. The high percentage means good compliance which means less AED skipping in a month.

CONTACTS AND LOCATIONS:
Overall Officials: Hunmin Kim, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea